CLINICAL TRIAL: NCT02644551
Title: The Efficacy of CELEXT07 in the Treatment of Toenail Onychomycosis: a Phase 2, Randomized, Double-blind Study
Brief Title: The Efficacy of CELEXT07 in the Treatment of Toenail Onychomycosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: 9305-9954 Quebec Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CELEXT07-01
Record Dates: First submitted 2015-12-29; First posted 2016-01-01 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — Ciclopirox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CELEXT07 (Experimental): suspension that is applied topically to the infected nail(s) daily.
  Interventions: Drug: CELEXT07
- placebo (Placebo Comparator): placebo is a suspension that simulates the physical properties of the experimental agent CELEXT07. It is applied topically to the infected nail(s) daily.
  Interventions: Other: vehicle solution
- Penlac (Active Comparator): Is a standard of care for the condition and is applied topically to the infected nail(s) daily.
  Interventions: Drug: Penlac

INTERVENTIONS:
Drug: CELEXT07
  Arms: CELEXT07
Drug: Penlac
  Other Names: topical Penlac nail lacquer
  Arms: Penlac
Other: vehicle solution
  Other Names: placebo
  Arms: placebo

SUMMARY:
This will be an interventional safety and efficacy study of CELENT07 when used as a topical treatment of onychomycosis in the toenails (tinea unguium) of adults 18 years and older. This is randomized, double-blind, parallel design, placebo and active controlled study in patients with mild to moderate toenail distal lateral subungual onychomycosis (DLSO) (n=120). Subjects will be randomized (1:1:1) to receive CELENXT07, placebo of CELENXT07 or PENLAC®, daily for 52 weeks. Efficacy assessments will include complete cure, mycologic cure and clinical efficacy and safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible to be included in the study only if they meet all of the following criteria:

1. Age > 18.
2. Clinically diagnosed onychomycosis of the target nail.
3. Presence of mild to moderate onychomycosis, defined as 20-50% of the area of the target nail being clinically affected.
4. Has a positive KOH examination from the target nail.
5. Has a positive dermatophyte culture from the target nail.
6. Written informed consent obtained.
7. Subject agreed to follow the protocol.

Exclusion Criteria

Subjects will be excluded from the study if they meet any of the following criteria:

1. Presence of any disease or condition that might cause nail abnormalities or may interfere with the evaluation of the study drug.
2. Use of any systemic antifungal therapy within 4 weeks prior to the Screening visit or non-responsive to systemic antifungal therapy for onychomycosis.
3. Use of any prescription or over-the-counter topical antifungal therapy for the toenails within 4 weeks prior to the Screening visit.
4. Woman who is pregnant, nursing an infant, or planning a pregnancy during the study period.
5. Inability to understand and comply with the instructions of the study
6. Patients less than age 18
7. Individuals with known allergy/hypersensitivity to Thuja occidentalis, Chelidonium majus, Eucalyptus citriodora, Tea tree or Thymus vulgaris.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy Assessed by Complete Cure Rate at the End of Study (Week 52) After Treating for 52 Weeks | week 52
  Complete cure is defined as negative KOH microscopy and negative culture for dermatophytes.
  and no residual involvement of the target toenail. The complete cure is a composite binary variable defined as "Yes" if:
  * Mycological cure (negative KOH and negative culture for dermatophytes) and
  * No residual involvement of the target toenail "No" if otherwise

SECONDARY OUTCOMES:
Efficacy Assessed by Clinical Efficacy at the End of Study After Treating Patients for 52 Weeks. | week 52
  Clinical effectiveness is defined as negative KOH microscopy and negative culture for dermatophytes and <= 10% residual involvement of the target toenail.Clinical effectiveness is a composite binary variable defined as "Yes" if
  * Mycological cure (negative KOH and negative culture for dermatophytes) and ◦= 10% residual involvement of the target toenail "No" if otherwise
Efficacy Assessed by Mycological Cure (Negative Culture and Negative KOH Microscopy) at the End of Study After Treating Patients for 52 Weeks. | week 52
  Mycological cure is defined as negative KOH microscopy and negative culture for dermatophytes.
  Mycological cure is a composite binary variable defined as "Yes"if :
  * Negative microscopy and
  * Negative culture for dermatophytes "No" if otherwise.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | week 52

CONTACTS AND LOCATIONS:
Overall Officials: Céline Devaux, MD, FRCPC, Principal Investigator — 9305-9954 Quebec Inc; Guy Chamberland, M.Sc., Ph.D., Study Director — 9305-9954 Quebec Inc
Locations (1):
- Clinique podiatrique de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided